CLINICAL TRIAL: NCT00558688
Title: A Photodynamic Therapy for Treatment of Actinic Keratoses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology-Head and Neck Surgery, and Surgery, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STU00000312
Record Dates: First submitted 2007-11-13; First posted 2007-11-15 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Photochemotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Light Therapy
  Interventions: Procedure: Photodynamic therapy
- 2 (Experimental): Light Therapy
  Interventions: Procedure: Photodynamic therapy

INTERVENTIONS:
Procedure: Photodynamic therapy — Photodynamic therapy applied to actinic keratoses

SUMMARY:
The purpose of this study is to compare the efficacy of photodynamic therapy with 5-aminolevulinic acid and intense pulsed light vs absence of treatment for actinic keratoses.

DETAILED DESCRIPTION:
This study seeks to evaluate the efficacy of photodynamic therapy with 5-aminolevulinic acid and intense pulsed light vs. absence of treatment for actinic keratoses

ELIGIBILITY:
Inclusion Criteria:

Age greater than or equal to 18 years

* Have a t least 4 nonhypertrophic AK lesions on the body
* The subjects are in good health
* The subject has the willingness and the ability to understand and provide informed consent for the use of their tissue and communicate to the investigator

Exclusion Criteria:

* Subjects who are pregnant or lactating
* Subjects with a history of cutaneous photosensitivity or porphyria, hypersensitivity to porphyrins, or photodermatosis
* Subjects with use of photosensitizing drugs within 1 week of study start
* Subjects with use of topical medications such as corticosteroids, alpha-hydroxyacids or retinoids 2 weeks before study entry
* Subjects with systemic steroid therapy within 4 weeks before study entry
* Subjects who received previous treatment of target AKs
* Subjects with systemic treatment with chemotherapeutic agents, masoprocol (Actinex), immunotherapy, or retinoids within 2 months of study entry
* Subjects with prior history of hypersensitivity reactions to lidocaine
* Subjects who are unable to understand the protocol or to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Visual assessment of lesions | 4 weeks

SECONDARY OUTCOMES:
Patient subjective assessment and Safety | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States